CLINICAL TRIAL: NCT05896852
Title: Healthy Lifestyles: A Home Based Physical Activity Intervention in Persons Living With HIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004962
Record Dates: First submitted 2023-05-11; First posted 2023-06-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Masking Description: N/A all study participants will be included in the intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will increase their physical activity over 6 months as tolerated,
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — Participants will increase their physical activity through walking.

SUMMARY:
This study is being done to understand how a physical activity walking intervention affects metabolic parameters (i.e., blood sugar, cholesterol, certain body measurements) in people with and without HIV. This study involves a physical activity intervention where participants will progressively increase activity as tolerated over a six month period.

DETAILED DESCRIPTION:
This study is being done to understand how a physical activity walking intervention affects metabolic parameters (i.e., blood sugar, cholesterol, certain body measurements) in people with and without HIV. This study involves a physical activity intervention where participants will progressively increase the total number of daily steps to approximately 10,000 steps/day as tolerated. We will monitor participant steps and physical activity using a physical activity monitor. The study will consist of 5 in-person study visits where participants will complete body measurements, laboratory testing (for metabolic parameters e.g. blood sugar and cholesterol), and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Persons living with or without HIV
* Metabolic Syndrome or risk factors for metabolic syndrome with BMI >=30
* Able to provide informed consent
* No physical limitations that prevent walking for more than 10 minutes
* Can provide evidence of medical clearance by healthcare provider, if required before or during the study

Exclusion Criteria:

* Currently exercising regularly (at least 2x weekly of at least 20minutes of moderate or vigorous activity)
* Current enrollment in another physician activity and/or dietary clinical trial or on diet/weight-loss program
* Active plans for bariatric surgery
* Inability to commit to the intervention schedule
* Not eligible as per screening form
* Currently pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Study Activities (Recruitment) | 6 months
  To determine acceptability of study activities investigators will determine overall recruitment and determine percentage of the target recruitment that enrolled in the study at the 6 month study completion point (goal = 90% of our target).
Acceptability of Study Activities (Attrition) | 6 months
  Investigators will measure attrition by determination of the number of participants who complete all study visits (measured by total number of participants who complete the baseline, 3-month, and 6-month study visits - goal >75%). These will be assessed at the end of the 6-month study period.
Adherence to Study Activities of Study Activities | 6 months
  Investigators will determine adherence to study activities by determination of the completion of study visits, completion of laboratory testing at study visits, and completion of step counting journals. Investigators will assess total number of documented study visits, completion of laboratory testing, and assessment of total number of days steps were entered in step logs. Investigators will assess the total number of visits, laboratory blood draws, and entries in to step log at each visit and determine overall percentage completed.

SECONDARY OUTCOMES:
Metabolic Parameters (Laboratory Measurement - blood glucose) | 6 months
  Laboratory measurements including fasting blood glucose (mg/dL) will be at baseline, 3-month, and 6-month visits. Change (increase/decrease) in the fasting blood glucose measurement will be assessed.
Metabolic Parameters (Laboratory Measurement - lipids) | 6 months
  Laboratory measurements including lipids (mg/dL) will be at baseline, 3-month, and 6-month visits. Change (increase/decrease) in the lipid measurements will be assessed.
Metabolic Parameters (Laboratory Measurement - HBA1c) | 6 months
  Laboratory measurements including HBA1c (mmol/mol) will be measured at baseline, 3-month, and 6-month visits. Change (increase/decrease) in the HBA1c measurement will be assessed.
Body Composition (Waist Circumference [cm]) | 6 months
  Body measurement including waist circumference in centimeters will be assessed at baseline, 3-month, and 6-month follow-up visits. Changes (increase/decrease) waist circumference will be assessed.
Body Composition (BMI [kg/m^2]) | 6 months
  Body measurement including BMI [kg/m^2] will be assessed at baseline, 3-month, and 6-month follow-up visits. Changes (increase/decrease) BMI will be assessed.
Quality of Life (Health-Related Quality of Life (SF-36)) | 6 months
  Health related quality of life will be assessed using the Health-Related Quality of Life (SF-36) scale. The scale includes eight measures - physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores range from 0 (worst) to 100 (best). Changes will be assessed from baseline to responses at the 6 month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No